CLINICAL TRIAL: NCT06016816
Title: The Effect of Bilateral Sphenopalatine Ganglion Block on Postoperative Pain in Patients to be Subject to Septorhinoplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTosunSoner
Record Dates: First submitted 2023-08-11; First posted 2023-08-30 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia of Mucous Membrane
Keywords: sphenopalatine ganglion block; septhorhinoplasty; general anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic bilateral sphenopalatine ganglion block (Active Comparator): After the induction of general anesthesia, one group (Group: 1) will be administered 8mg dexamethasone and 10mg bupivacaine submucosal,
  Interventions: Procedure: Bilateral endoscopic sphenopalatine ganglion block
- Placebo (Placebo Comparator): Placebo group (group:2) will be administered 4 cc saline. aspects will be evaluated.
  Interventions: Procedure: placebo

INTERVENTIONS:
Procedure: Bilateral endoscopic sphenopalatine ganglion block — After the induction of general anesthesia, one group (Group: 1) will be administered 8mg dexamethasone and 10mg bupivacaine submucosal,
  Arms: Endoscopic bilateral sphenopalatine ganglion block
Procedure: placebo — Placebo group (group:2) will be administered 4 cc saline. aspects will be evaluated.
  Arms: Placebo

SUMMARY:
The aim of this study is to examine the effects of bilateral sphenopalatine ganglion block on surgical conditions, hemodynamics, intraoperative and postoperative analgesic use, recovery characteristics, and postoperative pain during septorhinoplasty under general anesthesia. The study was planned as double-blind, randomized, controlled. 72 patients who will undergo septorhinoplasty surgery will be collected. (g power analysis was performed.) Evaluation of the effectiveness of bilateral sphenopalatine ganglion block was planned. Patients will be divided into 2 equal groups (36 patients). After the induction of general anesthesia, one group (Group: 1) will be administered 8mg dexamethasone and 10mg bupivacaine submucosal, the other group (group:2) will be administered 4 cc saline. aspects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

- patients with an ASA score of I-II and between the ages of 17-45 years, who were to undergo general anesthesia with desflurane, were included in the study.

Exclusion Criteria:

* Patients aged <17 and >45 years, patients with liver and/or kidney failure, obese patients (BMI >30), trauma patients, ASA III-IV patients, patients with bleeding disorders, those using drugs that may affect the coagulation system, patients with cardiomyopathy, cerebrovascular disease, immobility, and malnutrition were excluded from the study.

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | Postoperative 0-2 hours, 2-8 hours,8-24 hours
  They will be numbered from 1 to 10.
  1 mildest 10 most severe pain

SECONDARY OUTCOMES:
Riker Agitation Scale | Immediately after extubation
  7 Dangerous Agitation 6 Very Agitated 5 Agitated 4 Calm and Cooperative 3 sedated 2 Very Sedated A
  1 Unarousable
mean arterial pressure | when you come to the operating room table after anesthesia induction Intraoperative 30 minutes after extubation
  mmhg
heart rate | when you come to the operating room table after anesthesia induction Intraoperative 30 minutes after extubation
  beats\minute
intraoperative remifentanil consumption | intraoperative
  The intraoperative ultiva infusion dose was recorded to the patient.
edema questionnaire | Postoperative 0-2 hours, 2-8 hours,8-24 hours
  Periorbital edema was evaluated as present or absent questionnaire
hematoma questionnaire | Postoperative 0-2 hours, 2-8 hours,8-24 hours
  Hematoma was evaluated as present or absent questionnaire
vomiting questionnaire | Postoperative 0-2 hours, 2-8 hours,8-24 hours
  was evaluated as present or absent questionnaire
Oral analgesic use | In the first 24 hours after surgery
  Analgesic use in the first 24 hours was questioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Diyarbakır, Kayapınar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No